CLINICAL TRIAL: NCT02194114
Title: Dietary Protein Intake and Its Effect on Nitrogen Balance in Maintenance Hemodialysis (MHD) Patients
Brief Title: Dietary Protein Requirements in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10602
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Renal Failure; End-Stage Renal Disease
Keywords: Chronic Renal Failure; End-Stage Renal Disease; Nitrogen Balance; Dietary Protein Intake
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Protein Intake (Experimental): One treatment Arm; Protein Diet: All patients will be fed the following five diets, in random order, each for 17-19 days: 0.6 g protein/kg/day, 0.8 g protein/kg/day, 1.0 g protein/kg/day, 1.15 g protein/kg/day, 1.3 g protein/kg/day.
  Interventions: Other: Protein Diet

INTERVENTIONS:
Other: Protein Diet — Protein diets fed for 17-19 days to each patient in random order: 0.6 g protein/kg/day, 0.8 g protein/kg/day, 1.0 g protein/kg/day, 1.15 g protein/kg/day, 1.3 g protein/kg/day.

SUMMARY:
The primary purpose of this study is to assess dietary protein requirements in clinically stable maintenance hemodialysis (MHD) patients. It is hypothesized that the average dietary protein intake (DPI) that will maintain nitrogen balance is 1.00 g protein/kg/day, but that a safe intake that maintains balance in almost all MHD patients is about 1.25g protein/kg/day.

DETAILED DESCRIPTION:
A high proportion of maintenance hemodialysis (MHD) patients have protein-energy malnutrition (PEM) which is a powerful predictor of high morbidity and mortality. Although inflammation may contribute to PEM, low dietary protein intake (DPI) is often a contributing factor. The usual DPI of MHD patients in about 1.0 g protein/kg/day, whereas expert groups recommend = 1.20 g protein/kg/day. However, these recommendations are based upon few studies, often of insufficient duration, that were usually carried out with obsolete types of dialysis therapy.

We will examine the response to different levels of dietary protein intake (0.6-1.3 g protein/kg/day) under classical balance techniques with carefully controlled dietary intakes, living, conditions, and collection of nitrogen outputs and carefully measured nitrogen intakes and outputs.

ELIGIBILITY:
Inclusion Criteria:

* Ages from 30 years through 65 years
* Both men and women and all ethnic and racial groups
* Treatment with MHD for 6 months or greater
* Hemoglobin of at least 11 g/dL
* Neurological examination indicating no severe neuropathy
* A negative test for peripheral arterial occlusive disease

Exclusion Criteria:

* Obesity: body weight greater than >115% of standard
* History of active cancer other than basal cell carcinoma
* Symptomatic severe ischemic heart disease, uncontrolled serious dysrhythmias, uncontrolled congestive heart failure, poorly controlled hypertension, severe musculoskeletal disease, arthritis or amputations of the lower extremities
* Insulin dependent or insulin independent diabetes mellitus
* Severe lung or liver disease, uncontrolled asthma, active vasculitis. Severe chronic infection or any other acute or chronic inflammatory or catabolic illnesses
* Psychosis, inability to give informed consent, evidence that patient will not comply with study protocol
* Alcohol or other recreational drug abuse
* Patients who received L-carnitine or anabolic hormones within the previous 6 months
* Pregnancy
* Patients who are physically and/or psychologically incapable of undergoing the protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Nitrogen Balance | One year

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Kopple, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Derived] Shah A, Bross R, Shapiro BB, Morrison G, Kopple JD. Dietary energy requirements in relatively healthy maintenance hemodialysis patients estimated from long-term metabolic studies. Am J Clin Nutr. 2016 Mar;103(3):757-65. doi: 10.3945/ajcn.115.112995. Epub 2016 Feb 10. PMID 26864370